CLINICAL TRIAL: NCT00888966
Title: Evaluation of Oxidative Stress After Out of Hospital Cardiac Arrest Treated With Moderate Hypothermia
Brief Title: Oxidative Stress and Cardiac Arrest
Status: Completed | Type: Observational
Sponsor: Institut d'Anesthesiologie des Alpes Maritimes (Other)
Responsible Party: Orban MD, CHU de Nice
Other Study IDs: IAAM 2009-2
Record Dates: First submitted 2009-04-25; First posted 2009-04-28 (Estimated); Last update posted 2011-07-04 (Estimated); Status verified 2011-06

CONDITIONS: Heart Arrest
Keywords: heart arrest; oxidative stress; lactic acid; outcome
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Out of hospital cardiac arrest: Out of hospital cardiac patients successfully resuscitated and admitted to ICU

SUMMARY:
Cardiac arrest is a major health problem reaching 375000 cases in Europe each year. Only 5 to 31 % survive after an out of hospital cardiac arrest (OHCA). The main complication after OHCA is the anoxic encephalopathy. Recently mild hypothermia has shown a beneficial effect on survival. But the mechanisms underlying these therapy are not clear.

Cardiac arrest is an example of ischemia reperfusion of the entire body. And it is well demonstrated that reperfusion generates an oxidative stress. But it has never been shown in a clinical setting.

The aim of the study is to evaluate oxidative stress after out of hospital cardiac arrest treated with mild hypothermia.

ELIGIBILITY:
Inclusion Criteria:

* Out of hospital cardiac arrest

Exclusion Criteria:

* refractory shock
* moribund patient
* resuscitation > 60 minutes
* hypothermia < 30 degrees

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: community sample
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2006-04; Primary Completion 2010-06 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Oxidative stress markers and antioxidants after out of hospital cardiac arrest | 4 days

SECONDARY OUTCOMES:
Lactate after out of hospital cardiac arrest | 4 days
Outcome after out of hospital cardiac arrest | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Carole Ichai, MD, PhD, Study Chair — Centre Hospitalier Universitaire de Nice
Locations (1):
- CHU de Nice, Nice, France